CLINICAL TRIAL: NCT02909699
Title: Cardiovascular Health of Older Adults and Resveratrol
Brief Title: Cardiovascular Health of Older Adults and Resveratrol (CORE)
Acronym: CORE
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601756
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Aging
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dose 1: 1,000mg of resveratrol per day (1 pill 3 times per day). This ancillary study will be observational without drug administration.
  Interventions: Other: Observation
- Dose 2: 1,500mg of resveratrol per day (1 pill 3 times per day)
  Interventions: Other: Observation
- Placebo: Alike looking 1 pill 3 times per day
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — In this trial, cardiovascular function will be measured without drug administration. The drug will be administered within the main trial.

SUMMARY:
This study will investigate how resveratrol (phenol present in red grapes, wine and peanuts) can improve heart muscle function and ability of arteries to dilate in response to an increase in blood flow in adults 65 years of age and older. Additionally, investigators will look at how resveratrol can improve functioning of cells (cellular house-keeping) which can be related to cardiovascular function.

DETAILED DESCRIPTION:
Age-related declines in left ventricular function and endothelium-dependent vasodilation increase the risk for cardiovascular (CV) disease and premature death in older adults. Structural changes to the arterial wall and cardiac muscle are indicated as a cause and appear to be induced by age-related oxidative stress and inflammation and reduced levels of autophagy, the cellular "house-keeping system". Pre-clinical studies indicate that resveratrol (RSV), a polyphenol present mostly in grapes and red wine, may improve left ventricular cardiac muscle and endothelial vasodilator function. Although, RSV has been shown to induce autophagy and improve CV function in animals, evidence for its effects on the CV system in humans is lacking, and there is a need for clinical trials to better understand the effects of RSV on CV function in humans. Because older adults are most likely to have impairments in the central and peripheral CV systems, they represent an ideal population to test the effects of RSV on CV function. Therefore, the central hypothesis is that RSV supplementation will improve age-related left ventricular cardiac muscle function and arterial vasodilation in older adults (> 65 years). The participants will undergo 90 days of RSV treatment (n=12) (1,000mg/day), or (n=12) (1,500mg/day) or placebo (n=12). Before and after the intervention, investigators will non-invasively investigate left ventricular and arterial vasodilator function. Additionally, investigators will examine cardiac muscle damage and inflammatory biomarkers in blood and autophagy and endothelial function protein levels and in skeletal muscle to better understand molecular mechanisms that may underlie the hypothesized beneficial effects of RSV on cardiovascular health in older adults.

ELIGIBILITY:
Inclusion Criteria:

All the criteria are the same as in the parent R01 (IRB201400439). Participants must meet all inclusion criteria listed below in order to participate in this study.

* Ability to understand study procedures and to comply with them for the entire length of the study;
* Age 65 years and older;
* Moderately functioning (i.e. a summary score of 4 - 12 on the Short Physical Performance Battery);
* Body Mass Index (BMI) range: 20-39.9 kg/m2;
* Willingness to undergo all testing procedures.

Exclusion Criteria:

All candidates meeting any of the exclusion criteria listed below at baseline will be disqualified from study participation.

* Non-English speaking individual.
* Failure to provide informed consent;
* Allergy/sensitivity to grapes or Japanese knotweed;
* Current dietary supplementation of grape seed extract or ginko biloba;
* Consumption of ≥ 8 oz. of red wine/dealcoholized red wine/red or purple grape juice more than once weekly;
* Consumption of any dietary supplements containing resveratrol, quercetin, or P. cuspidatum in the previous 90 days;
* Active treatment for cancer, stroke (< 6 months), peripheral vascular disease, coronary artery disease, myocardial infarction (< 6 months), congestive heart failure (stage III or IV), valvular heart disease, major psychiatric disease, severe anemia (blood levels of Hemoglobin < 8 g/dl), bleeding disorders or other blood disorders, liver or renal disease, diabetes, severe osteoarthritis, blindness or deafness, fracture in upper or lower extremity ( < 6 months), upper or lower extremity amputation, or Parkinson's disease;
* Cognitive impairment (i.e. Mini Mental Status Exam ≤ 23 & Clinical Dementia Rating ≥1);
* History of significant head injury;
* Physical activity (i.e. running, bicycling, etc.) ≥ 150 min/week;
* Excessive alcohol use (> 2 drinks/day) or alcohol abuse (> 5 drinks/day for males, or > 4 drinks/day for females);
* History of substance abuse within the past six months;
* Mood disorder (i.e. Center for Epidemiological Studies - Depression (CES-D) ≥ 16);
* History of tobacco use within the past three years;
* Resting heart rate > 120 bpm at screening visit;
* Systolic blood pressure > 160 mm Hg at screening visit;
* Diastolic blood pressure > 90 mm Hg at screening visit;
* Fasting glucose ≥ 126 mg/dL at screening visit;
* Abnormalities in blood chemistry parameters, defined by blood chemistry marker outside of healthy range) as determined by study physician
* Current use of

  * anabolic treatments (e.g. growth hormone or testosterone),
  * anticholinesterase inhibitor (e.g. Aricept),
  * hormone replacement (e.g. Estrogen),
  * anticoagulant therapies (note: aspirin -anti-platelet use (≤ 81mg/day) is permitted) or
  * use of anti-inflammatory medications more than 3 times per week.;
* Participation in another non-observational clinical trial, or has received an investigational product within 30 days prior to screening/enrollment;
* Refuse to refrain from CoQ10 or alpha-lipoic acid while enrolled in the study.

Temporary Exclusion Criteria

A person meeting any of the following temporary exclusion criteria at the time of screening would not be enrolled but may be re-screened at a later date. A period of 4 weeks is the minimum amount of time required before re-screening for the following conditions can be done.

* Recent bacterial/viral infection (< 2 weeks);
* Acute febrile illness in past 2 months;
* High blood pressure (i.e. ≥ 140/90 mm Hg but ≤ 160/90) at the screening visit; Major surgery or hip/knee replacement (< 6 months);

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Moderately functioning older adults.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Speckle tracking analyses | Change from Baseline and 3 months
  Speckle tracking analyses will be performed using advanced quantification software version. Short axis and long axis images will be automatically divided into six segments. Automated tracking of myocardial speckles will be reviewed and manually adjusted as minimally as possible. The tracking quality of each segment will be visually evaluated and if tracking is felt to be inaccurate, strain analysis of that segment will not be included. Speckle tracking analysis provides peak and time to peak measures of circumferential, radial and longitudinal strain and strain rate in 18 left ventricle (LV) segments.

SECONDARY OUTCOMES:
Flow-mediated dilation | Change from baseline and 3 months
  A duplex ultrasound image of the brachial artery (i.e., 2-D image and spectral Doppler waveforms) will be obtained ∼7 cm proximal to the antecubital fossa.
Autophagy measured by Enzyme-linked immunosorbent assay (ELISA) | Baseline and 3 months
  Autophagy will be measured using Enzyme-linked immunosorbent assay (ELISA), a test that uses antibodies and color change to identify a substance.
Endothelin-1 protein expression will be measured by Western Blot | Change from baseline and 3 months
  Endothelin-1 protein expression will be measured using Western Blot which is used to identify specific amino-acid sequences in proteins.
Endothelial function endothelial nitric oxide synthase (eNOS) will be measured by Western Blot | Change from baseline and 3 months
  Endothelial function endothelial nitric oxide synthase will be measured using Western Blot which is used to identify specific amino-acid sequences in proteins.
Endothelin-1 protein expression will be measured by Enzyme-linked immunosorbent assay (ELISA) | Change from baseline and 3 months
  Endothelin-1 protein expression will be measured using Enzyme-linked immunosorbent assay (ELISA), a test that uses antibodies and color change to identify a substance.
Endothelial function endothelial nitric oxide synthase (eNOS) will be measured by Enzyme-linked immunosorbent assay (ELISA) | Change from baseline and 3 months
  Endothelial function endothelial nitric oxide synthase will be measured using Enzyme-linked immunosorbent assay (ELISA), a test that uses antibodies and color change to identify a substance.
Autophagy measured by Western Blot | Change from Baseline and 3 months
  Autophagy will be measured using Western Blot which is used to identify specific amino-acid sequences in proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Mankowski, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No